CLINICAL TRIAL: NCT02449226
Title: Accuracy of Point-of-Care Measurement of Electrolytes, Glucose, Hemoglobin and Hematocrit With the RapidPoint 500 Blood Gas Analyser
Brief Title: Accuracy of Point-of-Care Measurement With the RapidPoint 500 Blood Gas Analyser
Acronym: (POCREA)
Status: Completed | Type: Observational
Sponsor: Hôpital Européen Marseille (Other)
Responsible Party: Principal Investigator, Jerome Allardet-Servent, MD, M.D, M.Sc, Hôpital Européen Marseille
Other Study IDs: 2015-A00718-41
Record Dates: First submitted 2015-05-17; First posted 2015-05-20 (Estimated); Last update posted 2016-02-23 (Estimated); Status verified 2016-02

CONDITIONS: Critical Care; Electrolytes; Point-of-Care Systems

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
ICU patients are at high risk of ionic or metabolic disturbances during the course of their critical illness. Some of these disturbances might be life-threatening and require rapid response from physicians. Point-of-Care determination of electrolytes, glucose, hemoglobin and hematocrit ensures early detection (within 1 minute) of abnormal values and allows rapid and appropriate therapy. This technology has largely improved the quality of care in ICU. However, the accuracy of the measurement of those parameters had to be close enough to the reference method, usually perfomed in the central lab but time consuming. Recently, a novel generation of blood gas analyser has been released. Among them, the RapidPoint 500 is mounted with a 28-day cartridge which provides automatic calibrations and quality controls several times a day. Such a technology dramatically decreases the need for labs technical interventions. To date, there is no data reporting the accuracy of this device. Therefore, the investigators' aim is to compare the accuracy of the RapidPoint 500 with a reference measurement performed at the central laboratory (Beckman&Coulter AU5800 for electrolytes and Beckman&Coulter DXH for hemoglobin).

ELIGIBILITY:
Inclusion Criteria:

* Current stay in ICU
* Presence of an indwelling arterial catheter (radial or femoral)
* Prescription by physicians of a blood gas analysis and a laboratory analysis for the next morning

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients staying in our ICU and equipped with an indwelling arterial catheter for whom clinicians prescribe together an arterial blood gas analysis and a biological laboratory analysis.
  The study will take place over a 1 month period. A total of 300 pairs of samples is targeted.
Sampling Method: Non-Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2015-05; Primary Completion 2015-06 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
bias and limit of agreement | 1 month
  to describe the bias and limit of agreement between the tested method and the reference method for electrolytes, glucose, hemoglobin and hematocrit.
Dumming regression analysis | 1 month
  to describe the relation between the tested method and the reference method for electrolytes, glucose, hemoglobin and hematocrit.
Coefficient of correlation (Pearson) | 1 month
  to describe the correlation between the tested method and the reference method for electrolytes, glucose, hemoglobin and hematocrit.

CONTACTS AND LOCATIONS:
Overall Officials: Jérôme ALLARDET-SERVENT, MD, MSc, Principal Investigator — HOPITAL EUROPEEN MARSEILLE
Locations (1):
- Service de REANIMATION, HOPITAL EUROPEEN MARSEILLE, Marseille, France

REFERENCES:
- [Background] Ehrmeyer SS, Laessig RH, Leinweber JE, Oryall JJ. 1990 Medicare/CLIA final rules for proficiency testing: minimum intralaboratory performance characteristics (CV and bias) needed to pass. Clin Chem. 1990 Oct;36(10):1736-40. PMID 2170059
- [Background] Clinical and Laboratory Standards Institute (CLSI). Method Comparison and Bias Estimation Using Patient Samples; Approved Guideline-Third Edition. CLSI document EP9-A3 (ISBN 1-56238-887-8). Wayne, Pennsylvania, USA, 2013.